CLINICAL TRIAL: NCT04254159
Title: The Effects of Neuromuscular Electrical Stimulation to Muscle Strength, Functional Capacity and Quality of Life in Older Patients With Asthma: Randomized Controlled Trial
Brief Title: The Effects of Neuromuscular Electrical Stimulation in Older Patients With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Kadikoy Municipality Social Life Center (Unknown)
Responsible Party: Principal Investigator, Elif Develi, Physiotherapist, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ElifD
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Asthma
Keywords: Asthma; Neuromuscular Electrical Stimulation; Quadriceps Muscle Strength; Quality of Life
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Electrical Stimulation Group (Experimental): Asthma Education Aerobic Exercise Quadriceps Strengthening by superimposed NMES
  Interventions: Other: Superimposed Neuromuscular Electrical Stimulation; Behavioral: Patient Education Program; Other: Aerobic Exercise Training
- Control Group (Active Comparator): Asthma Education Aerobic Exercise Quadriceps Strengthening
  Interventions: Other: Quadriceps Strengthening; Behavioral: Patient Education Program; Other: Aerobic Exercise Training

INTERVENTIONS:
Other: Superimposed Neuromuscular Electrical Stimulation — NMES will be applied during each strengthening exercise session. A dual channel NMES stimulation device will be used with biphasic symmetric constant current impulses with a pulse width 300ms, a frequency of 50 Hz and a duty cycle of 10s on and 20s off protocol for 3 days a week for eight weeks.
  Arms: Neuromuscular Electrical Stimulation Group
Other: Quadriceps Strengthening — Quadriceps strength training will be done with resistive elastics bands for 3 days a week for eight weeks.
  Arms: Control Group
Behavioral: Patient Education Program — The aim of patient education is to increase awareness of patients about COPD and develop skills to better manage their disease. The patient education will be performed at least once via face to face interview. Education topics will be covered basic information about COPD, environmental risk factors, monitoring and managing the signs and symptoms of their disease, energy conservation techniques and relaxation positions to reduce dyspnea and usage of a specific inhaler.
Other: Aerobic Exercise Training — Exercise training will be comprised of cardiovascular endurance training with cycle ergometer and lower extremity strength training. The exercises will be done 3 days a week at the clinic under the supervision of physiotherapist. Total duration of exercise training will last for 8 weeks

SUMMARY:
The aim of the randomized controlled study is to investigate the effects of NMES superimposed on voluntary contraction combined with patient education and exercise training program in patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
When initial assessments will be completed, patients will be assigned to one of two possible sequences by simple randomization: Superimposed NMES group (SG) or control group (CG).

All volunteers will receive an COPD patient education program for once and conventional physiotherapy exercise program for COPD with the duration of 8 weeks. Additionally, superimposed NMES will be applied on quadriceps muscle of both limbs at the same time with voluntarily contraction of quadriceps muscle in SG.

All patients will be assessed in terms of functional capacity, pulmonary functions, quadriceps muscle endurance and strength, dyspnea, respiratory muscle strength and quality of life at the baseline and at the end of study. Data will be collected from all the patients at baseline and at the end of study (8 weeks) by the same physiotherapist who also will supervise the exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Having stable asthma
2. Participating to the study in a voluntary basis
3. Being 65 - 75 years old
4. Having 2 point or over score from "Modified Medical Research Council (MMRC)" Dyspnea Scale
5. Being motivated to participate and follow exercise program

Exclusion Criteria:

1. Having an asthma exacerbation in a last month
2. Other respiratory problems
3. Ischemic heart disease
4. Congestive heart disease
5. Pacemaker
6. Acute Cor Pulmonale
7. Neurological Diseases
8. Osteoporosis
9. Smoking

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Sit to Stand Test | 8 weeks
  Quadriceps muscle endurance will be evaluated with this test
Muscle Strength Test | 8 weeks
  Jtech Commander Power Track Muscle Testing Dynamometer, USA which quantifies muscle power will be used to assess the maximum voluntary contractions of quadriceps muscle in pound meter.
Six Minute Walking Test | 8 weeks
  Six-Minute Walking Test (6MWT) was used to evaluate functional capacity of volunteers.
Asthma Quality of Life Scale (AQOL) | 8 weeks
  Asthma quality of life questionnaire will utilize to assess quality of life of participants over two weeks prior to interview which is validated in Turkish population by Alpaydın et al.

SECONDARY OUTCOMES:
Modified Medical Research Council (MMRC) Dyspnea Scale | 8 weeks
  Perceived dyspnea which is any restrictions performing daily living activities will be measured by MMRC dyspnea scale.
Physical Activity Questionnaire for Elderly (PASE) | 8 weeks
  We will assess the physical activity status of the oler patients with asthma by using Physical Activity Questionnaire for Elderly (PASE).
Time Up and Go Test | 8 weeks
  Time Up and Go Test (TUG) will be used to evaluate the risk for falling in older patients with asthma.
Pulmonary Function Test | 8 weeks
  Medical International Research Spirodoc® Spiro, Italy brand named spirometry will be used to evaluate pulmonary functions of volunteers.
Respiratory Muscle Strength Testing | 8 weeks
  The Micro Medical Micro RPM, England respiratory pressure meter will be utilized to measure respiratory muscle strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Kadıköy Municipality Social Life Center, Istanbul, Kadıköy, Turkey (Türkiye)